CLINICAL TRIAL: NCT02935686
Title: A Randomized, Parallel-group, Placebo-controlled, Double-blind Phase 1/2a Study in Healthy HIV Uninfected Adults to Assess Safety/Tolerability and Immunogenicity of 2 Different Prime/Boost Regimens: Priming With Tetravalent Ad26.Mos4.HIV and Boosting With Tetravalent Ad26.Mos4.HIV and Either Clade C gp140 Plus Adjuvant OR a Combination of Mosaic and Clade C gp140 Plus Adjuvant
Brief Title: A Safety, Tolerability and Immunogenicity Study of 2 Different Regimens of Tetravalent Ad26.Mos4.HIV Prime Followed by Boost With Tetravalent Ad26.Mos4.HIV Along With Either Clade C gp140 Plus Adjuvant OR With a Combination of Mosaic and Clade C gp140 Plus Adjuvant in Healthy HIV Uninfected Adults
Acronym: IPCAVD-012
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108207; VAC89220HPX2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Results first posted 2025-01-07 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Ad26.Mos4.HIV + Clade C gp140 (Experimental): Participants will receive Ad26.Mos4.HIV vaccine at Week 0 and 12, followed by Ad26.Mos4.HIV vaccine + Clade C glycoprotein 140 vaccine containing 250 microgram (mcg) of total protein mixed with adjuvant (aluminium phosphate) at Week 24 and 48. Participants who receive all 4 vaccinations and are negative for HIV infection at Week 72 can consent to be included in a long-term extension (LTE) phase (approximately 3 years after Week 72).
  Interventions: Biological: Ad26.Mos4.HIV; Biological: Clade C gp140 plus adjuvant
- Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 (Experimental): Participants will receive Ad26.Mos4.HIV vaccine at Week 0 and 12; followed by Ad26.Mos4.HIV vaccine + combination of 125 mcg Mosaic gp140 and 125 mcg Clade C gp140 mixed with adjuvant (aluminum phosphate) at Week 24 and 48. Participants who receive all 4 vaccinations and are negative for HIV infection at Week 72 can consent to be included in a long-term extension (LTE) phase (approximately 3 years after Week 72).
  Interventions: Biological: Ad26.Mos4.HIV; Biological: Clade C gp140/Mosaic gp140 plus adjuvant
- Group 3: Placebo (Placebo Comparator): Participants will receive a single placebo injection at Weeks 0 and 12, followed by two placebo injections at Weeks 24 and 48.
  Interventions: Other: Placebo
- Group 1b: Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine (Experimental): Participants enrolled in the LTE phase will receive late boost vaccination Ad26.Mos4.HIV and bivalent gp140 within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, approximately 3 years after the 4th vaccination of the primary vaccination series).
  Interventions: Biological: Ad26.Mos4.HIV; Biological: gp140 HIV Bivalent Vaccine
- Group 2b: Placebo (Placebo Comparator): Participants will receive placebo injection at Week 192 -4 weeks/+4 months, that is, approximately 3 years after the 4th vaccination of the primary vaccination series.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ad26.Mos4.HIV — Ad26.Mos4.HIV at a dose of 5*10^10 viral particles (vp), administered intramuscularly.
  Arms: Group 1: Ad26.Mos4.HIV + Clade C gp140; Group 1b: Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine; Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Biological: Clade C gp140 plus adjuvant — Clade C gp140 vaccine containing 250 mcg of total protein, mixed with aluminum phosphate adjuvant, per 0.5 milliliter (mL) injection administered intramuscularly.
  Arms: Group 1: Ad26.Mos4.HIV + Clade C gp140
Biological: Clade C gp140/Mosaic gp140 plus adjuvant — Clade C gp140 and Mosaic gp140 (each 125 mcg of total protein) mixed with aluminum phosphate adjuvant, per 0.5 milliliter (mL) injection, administered intramuscularly.
  Arms: Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Other: Placebo — Placebo Containing 0.9 percent normal saline, administered intramuscularly.
  Arms: Group 2b: Placebo; Group 3: Placebo
Biological: gp140 HIV Bivalent Vaccine — gp140 HIV Bivalent Vaccine is adjuvanted protein co-formulation with a dosage strength of 80 mcg Clade C protein, 75 mcg Mosaic protein and 425 mcg aluminum (as aluminum phosphate adjuvant).
  Arms: Group 1b: Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine

SUMMARY:
The primary purpose of this study is to assess safety/tolerability of the different vaccine regimens and of a late boost vaccination; and to assess envelope (Env)-binding antibody (Ab) responses of the 2 different vaccine regimens.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), double-blind (neither physician nor participant knows the treatment received), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), parallel-group (each treatment group will be treated at the same time), multicenter (more than one clinical site) study in healthy human immunodeficiency virus (HIV)-uninfected adults. The main study will be conducted in 3 phases: a 6-week screening period; a 48-week vaccination period; and a follow-up period to the final main study visit at Week 72. A Long-term Extension (LTE) phase (approximately 3 years after Week 72) will be performed for participants randomized to Group 1 or Group 2, who receive all 4 vaccinations and are negative for HIV infection at Week 72. The approximate duration of the study will be approximately 78 weeks for participants not participating in the LTE phase and approximately 222 weeks for participants participating in the LTE phase but not receiving a late boost vaccination and approximately 246 (12-month follow-up) or 294 (24-month follow-up) weeks for participants receiving a late boost vaccination. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of medical history, physical examination, and vital signs measurement performed at screening
* Participants are negative for human immunodeficiency virus (HIV) infection at screening
* Participants are amenable to HIV-risk reduction counseling and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* All female participants of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at the screening visit, and a negative urine pregnancy test pre-dose on Day 1
* Participants are willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures
* Participant must be enrolled in the LTE phase to receive the late boost vaccination

Exclusion Criteria:

* Has chronic hepatitis B (measured by hepatitis B surface antigen test) or active hepatitis C (measured by hepatitis C virus [HCV] Ab test; if positive, HCV ribonucleic acid [RNA] polymerase chain reaction (PCR) test will be used to confirm active versus past HCV infection), active syphilis infection, chlamydia, gonorrhea, or trichomonas
* In the 12 months prior to randomization, participant has a history of newly acquired herpes simplex virus type 2 (HSV-2), syphilis, gonorrhea, non-gonococcal urethritis, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranulomavenereum, chancroid, or hepatitis B
* Participant has had major surgery (eg, requiring general anesthesia) within the 4 weeks before screening, or will not have fully recovered from surgery, or has surgery planned through the course of the study
* Participant has had a thyroidectomy or active thyroid disease requiring medication during the last 12 months (not excluded: a stable thyroid supplementation)
* Current or past drug/alcohol use that investigator assesses poses any more than a remotely increased risk of the ability of the participant to comply with the protocol requirements
* Has been in receipt of any licensed vaccine within 14 days prior to the first dose of study vaccine or placebo, plans to receive within 14 days after the first study vaccination, or plans to receive within 14 days before or after the second, third or fourth vaccination
* Is a recipient of a prophylactic or therapeutic HIV vaccine candidate at any time, or a recipient of other experimental vaccine(s) within the last 12 months prior to the Day 1 visit (Vaccination 1). For participants who received an experimental vaccine (except HIV vaccine) more than 12 months prior to the Day 1 visit (Vaccination 1), documentation of the identity of the experimental vaccine must be provided to the sponsor, who will determine eligibility on a case-by-case basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (13):
- United States (11):
  - Alabama Vaccine Research Clinic at UAB, Birmingham, Alabama
  - Bridge HIV, San Francisco, California
  - The Hope Clinic at Emory University, Decatur, Georgia
  - Brigham And Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Fenway Health, Boston, Massachusetts
  - Columbia University HIV Vaccine Unit, New York, New York
  - New York Blood Center, New York, New York
  - Strong Memorial Infectious Disease, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Seattle Vaccine Trials Unit, Seattle, Washington
- Walter Reed Project Clinical Research Center, Kericho, Kenya
- Center for Family Health Research/Project San Francisco, Kigali, Rwanda

REFERENCES:
- [Derived] Stieh DJ, Barouch DH, Comeaux C, Sarnecki M, Stephenson KE, Walsh SR, Sawant S, Heptinstall J, Tomaras GD, Kublin JG, McElrath MJ, Cohen KW, De Rosa SC, Alter G, Ferrari G, Montefiori D, Mann P, Nijs S, Callewaert K, Goepfert PA, Edupuganti S, Karita E, Seaman MS, Corey L, Baden LR, Pau MG, Schuitemaker H, Tomaka F; ASCENT/HVTN118/HPX2003 Study Team. Safety and Immunogenicity of Ad26-Vectored HIV Vaccine With Mosaic Immunogens and a Novel Mosaic Envelope Protein in HIV-Uninfected Adults: A Phase 1/2a Study. J Infect Dis. 2023 Apr 18;227(8):939-950. doi: 10.1093/infdis/jiac445. PMID 36348617

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From Week 192 (-4 weeks/+ 4 months), eligible and consenting participants in long-term extension (LTE) phase received late boost vaccination and continued in late boost vaccination phase. Hence, there is an overlap in the duration of LTE and late boost vaccination phase.
Groups:
- Group 1 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140: Participants in the main study received single intramuscular (IM) injection of Ad26.Mos4.HIV vaccine 5*10^10 viral particles (vp) at Weeks 0 and 12 (- 1 week/ + 3 weeks), followed by Ad26.Mos4.HIV vaccine 5*10^10 vp + Clade C glycoprotein 140 vaccine containing 250 micrograms (mcg) of total protein mixed with adjuvant (aluminum phosphate) IM injection at Weeks 24 (- 1 week/ + 3 weeks) and 48 (- 1 week/ + 3 weeks). Participants who received all 4 vaccinations and were negative for HIV infection at Week 72 and consented separately for an optional long-term extension (LTE) phase after Week 72 and were followed up until Week 216 (for participants who did not enter late boost vaccination phase) and up to any day between Week 188 to Week 208 for those who entered late boost vaccination phase.
- Group 2 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140: Participants in the main study received single IM injection of Ad26.Mos4.HIV vaccine 5*10^10 vp at Weeks 0 and 12 (- 1 week/ + 3 weeks), followed by Ad26.Mos4.HIV vaccine 5*10^10 vp + combination of Mosaic gp140 and Clade C gp140 containing 125 micrograms (mcg) of Clade C gp140 and 125 mcg Mosaic gp140 mixed with adjuvant (aluminum phosphate) IM injection at Weeks 24 (- 1 week/ + 3 weeks) and 48 (- 1 week/ + 3 weeks). Participants who received all 4 vaccinations and were negative for HIV infection at Week 72 consented separately for an optional long-term extension (LTE) phase after Week 72 and were followed up until Week 216 (for participants who did not enter late boost vaccination phase) and up to any day between Week 188 to Week 208 for those who entered late boost vaccination phase.
- Group 3 Main Study: Placebo: Participants received a single IM injection of placebo matching to Ad26.Mos4.HIV at Weeks 0 and 12 (- 1 week/ + 3 weeks), followed by placebo injections matching to AD26.Mos4.HIV and matching to Clade C + Mosaic gp140 at Weeks 24 (- 1 week/ + 3 weeks) and 48 (- 1 week/ + 3 weeks).
- Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine: Participants from Group 1 and 2 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with Ad26.Mos4.HIV and bivalent gp140 containing adjuvanted protein co-formulation with 80 mcg Clade C protein, 75 mcg Mosaic protein and 425 mcg aluminum (as aluminum phosphate adjuvant) as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
- Group 2b: LTE Then Late-boost Placebo: Participants from Group 1 and 2 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with placebo matching to Ad26.Mos4.HIV and matching to gp140 HIV bivalent as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
Period: Main Study (Week 0 up to Week 72)
Arm/Group | Group 1 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 | Group 2 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3 Main Study: Placebo | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Started | 26 | 103 | 26 | 0 | 0
Vaccinated | 26 | 100 | 26 | 0 | 0
Completed | 19 | 87 | 24 | 0 | 0
Not Completed | 7 | 16 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 9 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0
Not completed — Randomized but not vaccinated | 0 | 3 | 0 | 0 | 0
Period: Long-term Extension (Week 72 - 216)
Arm/Group | Group 1 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 | Group 2 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3 Main Study: Placebo | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Started | 14 | 76 | 0 | 0 | 0
Participants Entering LTE and Did Not Receive Late-boost (Weeks 72-216) | 3 | 33 | 0 | 0 | 0
Completed | 12 | 63 | 0 | 0 | 0
Not Completed | 2 | 13 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 8 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Period: Late Boost Vaccination (Week 192 - 288)
Arm/Group | Group 1 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 | Group 2 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3 Main Study: Placebo | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Started (Participants from LTE who received late-boost vaccination from Week 192 (-4 weeks/+ 4 months)) | 0 | 0 | 0 | 41 | 13
Completed | 0 | 0 | 0 | 39 | 11
Not Completed | 0 | 0 | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FA) consisted of all participants who were randomized and who received at least one dose of study vaccine.
Groups:
- Group 1: Ad26.Mos4.HIV + Clade C gp140: Participants in the main study received single intramuscular (IM) injection of Ad26.Mos4.HIV vaccine 5*10^10 viral particles (vp) at Weeks 0 and 12 (- 1 week/ + 3 weeks), followed by Ad26.Mos4.HIV vaccine 5*10^10 vp + Clade C glycoprotein 140 vaccine containing 250 micrograms (mcg) of total protein mixed with adjuvant (aluminum phosphate) IM injection at Weeks 24 (- 1 week/ + 3 weeks) and 48 (- 1 week/ + 3 weeks). Participants who received all 4 vaccinations and were negative for HIV infection at Week 72 and consented separately for an optional long-term extension (LTE) phase after Week 72 and were followed up until Week 216 (for participants who did not enter late boost vaccination phase) and up to any day between Week 188 to Week 208 for those who entered late boost vaccination phase.
- Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140: Participants in the main study received single IM injection of Ad26.Mos4.HIV vaccine 5*10^10 vp at Weeks 0 and 12 (- 1 week/ + 3 weeks), followed by Ad26.Mos4.HIV vaccine 5*10^10 vp + combination of Mosaic gp140 and Clade C gp140 containing 125 micrograms (mcg) of Clade C gp140 and 125 mcg Mosaic gp140 mixed with adjuvant (aluminum phosphate) IM injection at Weeks 24 (- 1 week/ + 3 weeks) and 48 (- 1 week/ + 3 weeks). Participants who received all 4 vaccinations and were negative for HIV infection at Week 72 consented separately for an optional long-term extension (LTE) phase after Week 72 and were followed up until Week 216 (for participants who did not enter late boost vaccination phase) and up to any day between Week 188 to Week 208 for those who entered late boost vaccination phase.
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3 Main Study: Placebo | Total
Number analyzed (Participants) | 26 | 100 | 26 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (7.07) | 31.8 (8.09) | 30.7 (10.11) | 31.1 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 59 | 15 | 90
  Male | 10 | 41 | 11 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 4 | 12
  Not Hispanic or Latino | 24 | 92 | 22 | 138
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 7 | 2 | 11
  Black or African American | 10 | 38 | 9 | 57
  White | 12 | 47 | 12 | 71
  Other | 2 | 8 | 3 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  KENYA | 1 | 4 | 0 | 5
  RWANDA | 7 | 26 | 7 | 40
  UNITED STATES | 18 | 70 | 19 | 107

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) for 7 Days Post-vaccination 1
Description: Number of participants with solicited local and systemic AEs for 7 days post-vaccination 1 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Solicited AEs were precisely local and systemic events for which the participant is specifically questioned and symptoms of which were noted by participant in their diary. Solicited local AEs included injection site pain/tenderness, erythema, and swelling/induration at the study vaccine injection site. Solicited systemic AEs included fever (temperature measurement), fatigue, headache, nausea, myalgia, and chills.
Time Frame: Up to 7 days post-vaccination 1 on Day 1 (up to Day 8)
Population: Full analysis set (FAS) included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- Group 3: Placebo: Participants received a single IM injection of placebo matching to Ad26.Mos4.HIV at Weeks 0 and 12 (- 1 week/ + 3 weeks), followed by placebo injections matching to AD26.Mos4.HIV and matching to Clade C + Mosaic gp140 at Weeks 24 (- 1 week/ + 3 weeks) and 48 (- 1 week/ + 3 weeks).
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 26 | 100 | 26
Participants
  Solicited local AE | 21 | 78 | 6
  Solicited systemic AE | 20 | 80 | 16

2. Primary Outcome: Main Study: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) for 7 Days Post-vaccination 2
Description: Number of participants with solicited local and systemic AEs for 7 days post-vaccination 2 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Solicited AEs were precisely local and systemic events for which the participant is specifically questioned and symptoms of which were noted by participant in their diary. Solicited local AEs included injection site pain/tenderness, erythema, and swelling/induration at the study vaccine injection site. Solicited systemic AEs included fever (temperature measurement), fatigue, headache, nausea, myalgia, and chills.
Time Frame: Up to 7 days post vaccination 2 (up to any day from Day 78 to Day 113) (vaccination 2 ranged from Day 78 to 106)
Population: FAS included all participants who were randomized and who received at least one dose of study vaccine. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 24 | 98 | 25
Participants
  Solicited local AE | 19 | 66 | 5
  Solicited systemic AE | 15 | 58 | 13

3. Primary Outcome: Main Study: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) for 7 Days Post-vaccination 3
Description: Number of participants with solicited local and systemic AEs for 7 days post-vaccination 3 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Solicited AEs were precisely local and systemic events for which the participant is specifically questioned and symptoms of which were noted by participant in their diary. Solicited local AEs included injection site pain/tenderness, erythema, and swelling/induration at the study vaccine injection site. Solicited systemic AEs included fever (temperature measurement), fatigue, headache, nausea, myalgia, and chills.
Time Frame: Up to 7 days post vaccination 3 (up to any day from Day 162 to Day 197) (vaccination 3 ranged from Day 162 to 190)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 23 | 92 | 25
Participants
  Solicited local AE | 18 | 73 | 12
  Solicited systemic AE | 10 | 55 | 8

4. Primary Outcome: Main Study: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) for 7 Days Post-vaccination 4
Description: Number of participants with solicited local and systemic AEs for 7 days post-vaccination 4 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Solicited AEs were precisely local and systemic events for which the participant is specifically questioned and symptoms of which were noted by participant in their diary. Solicited local AEs included injection site pain/tenderness, erythema, and swelling/induration at the study vaccine injection site. Solicited systemic AEs included fever (temperature measurement), fatigue, headache, nausea, myalgia, and chills.
Time Frame: Up to 7 days post vaccination 4 (up to any day from Day 330 to Day 365) (vaccination 4 ranged from Day 330 to 358)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 19 | 88 | 24
Participants
  Solicited local AE | 13 | 70 | 7
  Solicited systemic AE | 11 | 53 | 6

5. Primary Outcome: Main Study: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days Post-vaccination 1
Description: Number of participants with unsolicited AEs for 28 days post-vaccination 1 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to 28 days post-vaccination 1 on Day 1 (Up to Day 29)
Population: FAS included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 26 | 100 | 26
Participants | 8 | 40 | 12

6. Primary Outcome: Main Study: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days Post-vaccination 2
Description: Number of participants with unsolicited AEs for 28 days post-vaccination 2 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to 28 days post vaccination 2 (up to any day from Day 78 to Day 134) (vaccination 2 ranged from Day 78 to 106)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 24 | 98 | 25
Participants | 6 | 35 | 7

7. Primary Outcome: Main Study: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days Post-vaccination 3
Description: Number of participants with unsolicited AEs for 28 days post-vaccination 3 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to 28 days post vaccination 3 (up to any day from Day 162 to Day 218) (vaccination 3 ranged from Day 162 to 190)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 23 | 92 | 25
Participants | 5 | 38 | 8

8. Primary Outcome: Main Study: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days Post-vaccination 4
Description: Number of participants with unsolicited AEs for 28 days post-vaccination 4 were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to 28 days post vaccination 4 (up to any day from Day 330 to Day 358) (vaccination 4 ranged from Day 330 to 358)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 19 | 88 | 24
Participants | 3 | 30 | 5

9. Primary Outcome: Main Study: Number of Participants Who Discontinued Study Vaccination Due to AEs
Description: Number of participants who discontinued study vaccination due to AEs were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment.
Time Frame: From Baseline (Day 1) up to Week 72
Population: FAS included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 26 | 100 | 26
Participants | 1 | 0 | 0

10. Primary Outcome: Main Study: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with SAEs were reported. An AE was any untoward medical occurrence in a clinical study administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: From Baseline (Day 1) up to Week 72
Population: FAS included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 26 | 100 | 26
Participants | 0 | 0 | 0

11. Primary Outcome: Main Study and LTE Study: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Number of participants with adverse events of special interest (AESIs) were reported. As planned, confirmed HIV infection was the only event assessed as an AESI. AESIs (including potential AESIs) are significant AEs that are judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. AESIs (including potential AESIs) must be reported to the sponsor within 24 hours of awareness irrespective of seriousness (that is, serious and nonserious AEs) or causality.
Time Frame: From Baseline (Day 1) up to Week 216
Population: FAS: all participants who were randomized and received at least 1 dose of study vaccine in main study and continued in LTE and did not enter late boost vaccination phase. Due to change in planned analysis, safety data for main study and LTE were combined for Groups 1 and 2 as LTE was a follow-up for participants who were in main study in Groups 1 and 2; no intervention was given in LTE. As both phases involved same participants in continued monitoring, data reflects ongoing safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3 Main Study: Placebo
Number analyzed (Participants) | 26 | 100 | 26
Participants | 0 | 0 | 0

12. Primary Outcome: Late-boost (LB) Vaccination Phase: Number of Participants Who Discontinued Study Due to AEs
Description: Number of participants who discontinued study due to AEs were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment.
Time Frame: From Week 188 up to end of study (Week 288)
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 41 | 13
Participants | 0 | 1

13. Primary Outcome: Late-boost (LB) Vaccination Phase: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) for 7 Days Post Late Boost Vaccination
Description: Number of participants with solicited local and systemic AEs for 7 days post late boost vaccination were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Solicited AEs were precisely local and systemic events for which the participant is specifically questioned and symptoms of which were noted by participant in their diary. Solicited local AEs included injection site pain/tenderness, erythema, and swelling/induration at the study vaccine injection site. Solicited systemic AEs included fever (temperature measurement), fatigue, headache, nausea, myalgia, and chills.
Time Frame: Up to 7 days post late boost vaccination (up to any day from Day 1317 to Day 1464) (late boost vaccination ranged from Day 1317 to 1457)
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 41 | 13
Participants | 37 | 9

14. Primary Outcome: Late-boost (LB) Vaccination Phase: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days Post Late Boost Vaccination
Description: Number of participants with unsolicited AEs for 28 post late boost vaccination were reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to 28 days post late boost vaccination (up to any day from Day 1317 to Day 1485) (late boost vaccination ranged from Day 1317 to 1457)
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 41 | 13
Participants | 11 | 4

15. Primary Outcome: Late-boost (LB) Vaccination Phase: Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 10
Time Frame: From Week 188 up to end of study (Week 288)
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 41 | 13
Participants | 1 | 1

16. Primary Outcome: Late-boost (LB) Vaccination Phase: Number of Participants With AESIs of HIV Infection Up to End of Study
Description: Number of participants with AESIs up to the end of the study were reported. An AE was any untoward medical occurrence in a clinical study administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. AESIs (including potential AESIs) are significant AEs that are judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. AESIs (including potential AESIs) must be reported to the sponsor within 24 hours of awareness irrespective of seriousness (i.e, serious and nonserious AEs) or causality. Confirmed HIV infection was considered an AESI.
Time Frame: From Week 188 up to end of study (Week 288)
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 41 | 13
Participants | 0 | 2

17. Primary Outcome: Late-boost (LB) Vaccination Phase: Number of Participants With AESIs of Thrombosis With Thrombocytopenia Syndrome (TTS)
Description: Number of participants with AESIs of TTS were reported. An AE was any untoward medical occurrence in a clinical study administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. AESIs are significant AEs that are judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. AESIs must be reported to the sponsor within 24 hours of awareness irrespective of seriousness (i.e, serious and nonserious AEs) or causality. Thrombotic events and/or thrombocytopenia were considered as AESIs.
Time Frame: Up to 6 months post late boost vaccination (up to any day from Day 1317 to Day 1639) (late boost vaccination ranged from Day 1317 to 1457)
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 41 | 13
Participants | 0 | 0

18. Primary Outcome: Main Study: Geometric Mean of Envelope (Env) Clade A (92UG037.1), B (1990a), C (Con C), (C97ZA.012), Mos 1 Specific Binding Antibodies (Abs) Responses As Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 28
Description: Geometric mean of Env Clade A (92UG037.1), B (1990a), C (Con C), (C97ZA.012), Mos 1 specific binding Abs responses were assessed using ELISA.
Time Frame: Week 28
Population: PPI set included participants who received at least first 3 vaccines, as per protocol, had at least one measured post dose blood sample collected and were not diagnosed with HIV during study. Samples taken post Week 48 from participants in PPI set who missed or did not receive 4th vaccine in protocol specified time window (+/- 2 weeks) were excluded from analysis. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 20 | 90 | 25
ELISA units/milliliter (EU/mL)
  Clade A (92UG037.1) | 99731.9 [61923.3 to 160625.5] | 88412.7 [7592.1 to 102917.5] | 312.5 [312.5 to 312.5]
  Clade B (1990a) | 67190.3 [42923 to 105177.6] | 71067.3 [60104.7 to 84029.4] | 94.4 [71.8 to 123.9]
  Clade C (Con C) | 149924.9 [91195.3 to 246476.1] | 130235.2 [110383.5 to 153656.9] | 333.3 [303.9 to 365.5]
  Clade C (C97ZA.012) | 65644.1 [43866.4 to 98233.5] | 54942.6 [46038 to 65569.4] | 98.4 [70.7 to 136.9]
  Mos 1 | 69234.2 [40940.5 to 117081.3] | 73780 [60679.2 to 89709.3] | 39.1 [39.1 to 39.1]

19. Primary Outcome: Main Study: Geometric Mean of Envelope (Env) Clade A (92UG037.1), B (1990a), C (Con C), (C97ZA.012), Mos 1 Specific Binding Antibodies (Abs) Responses As Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 52
Description: as for outcome 18
Time Frame: Week 52
Population: PPI set was used in this analysis. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 17 | 82 | 23
ELISA units/milliliter (EU/mL)
  Clade A (92UG037.1) | 104042.2 [78120.7 to 138564.8] | 139725.1 [117861.4 to 165644.6] | 312.5 [312.5 to 312.5]
  Clade B (1990a): number analyzed (Participants) | 17 | 81 | 23
  Clade B (1990a) | 77042.3 [51359.9 to 115567.2] | 133424.3 [111903.8 to 159083.5] | 94.3 [72 to 123.5]
  Clade C (Con C) | 155117.3 [107852.7 to 223094.6] | 237501.1 [197847.5 to 285102.3] | 323.1 [301.5 to 346.2]
  Clade C (C97ZA.012) | 92936.2 [60391.6 to 143018.7] | 110083.7 [92455 to 131073.8] | 78.1 [78.1 to 78.1]
  Mos 1: number analyzed (Participants) | 15 | 82 | 23
  Mos 1 | 79595 [49206 to 128751.7] | 137520.1 [115722.2 to 163423.8] | 39.1 [39.1 to 39.1]

20. Primary Outcome: Main Study: Geometric Mean of Envelope (Env) Clade A (92UG037.1) B (1990a), C (Con C), (C97ZA.012), Mos 1 Specific Binding Antibodies (Abs) Responses As Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 72
Description: Geometric mean of Env Clade A (92UG037.1) B (1990a), C (Con C), (C97ZA.012), Mos 1 specific binding Abs responses were assessed using ELISA.
Time Frame: Week 72
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 17 | 84 | 21
ELISA units/milliliter (EU/mL)
  Clade A (92UG037.1) | 33049.4 [22287.3 to 49008.4] | 39174.4 [32083 to 47833.2] | 312.5 [312.5 to 312.5]
  Clade B (1990a) | 20625 [14107.1 to 30154.3] | 33177.5 [27444.9 to 40107.6] | 99.1 [69.7 to 140.8]
  Clade C (Con C): number analyzed (Participants) | 17 | 83 | 21
  Clade C (Con C) | 44505.6 [31448.4 to 62984.1] | 57596.5 [47597.1 to 69696.7] | 342 [300.4 to 389.4]
  Clade C (C97ZA.012) | 18236.1 [11989.7 to 27736.7] | 18857.2 [15759.6 to 22563.7] | 83.1 [73 to 94.6]
  Mos 1 | 16861.6 [11096.6 to 25621.5] | 25161.6 [20879.1 to 30322.6] | 40.9 [37.2 to 44.9]

21. Primary Outcome: Main Study: Percentage of Responders for Envelope (Env)-Specific Binding Antibody Titers at Week 28
Description: Percentage of responders for envelop (Env) Clade B (SC42261), Clade C (CH505TF), Clade A (9004S), Clade B (RHPA), Clade B (WITO), Clade C (1086C), Clade C (BF1266), CladeAE (conAE), Clade M(Con S)-specific binding antibody titers assessed using enzyme-linked immunosorbent assay (ELISA) were reported. The response was defined as post-baseline value greater than (>) lower limit of quantification (LLOQ) if baseline value less than (<) LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline value greater than or equal to (>=) LLOQ.
Time Frame: Week 28
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 19 | 82 | 22
percentage of responders
  Clade B (SC42261) | 100 [82.4 to 100] | 100.0 [95.6 to 100.0] | 0 [0 to 0]
  Clade C (CH505TF) | 100 [82.4 to 100] | 100 [95.6 to 100] | 0 [0 to 0]
  Clade A (9004S) | 100 [82.4 to 100] | 100 [95.6 to 100] | 0 [0 to 0]
  Clade B (RHPA) | 100 [82.4 to 100] | 100 [95.6 to 100] | 0 [0 to 0]
  Clade B (WITO) | 100 [82.4 to 100] | 100 [95.6 to 100] | 0 [0 to 0]
  Clade C (1086C) | 100 [82.4 to 100] | 100 [95.6 to 100] | 0 [0 to 0]
  Clade C (BF1266) | 100 [82.4 to 100] | 100 [95.6 to 100] | 0 [0 to 0]
  CladeAE (conAE) | 100 [82.4 to 100] | 100 [95.6 to 100] | 0 [0 to 0]
  Clade M(Con S) | 100 [82.4 to 100] | 100 [95.6 to 100] | 0 [0 to 0]

22. Primary Outcome: Main Study: Percentage of Responders for Envelope (Env)-Specific Binding Antibody Titers at Week 52
Description: as for outcome 21
Time Frame: Week 52
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 19 | 82 | 22
percentage of responders
  Clade B (SC42261) | 100 [78.2 to 100] | 100.0 [95.2 to 100.0] | 0 [0 to 0]
  Clade C (CH505TF) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]
  Clade A (9004S) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]
  Clade B (RHPA) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]
  Clade B (WITO) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]
  Clade C (1086C) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]
  Clade C (BF1266) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]
  CladeAE (conAE) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]
  Clade M(Con S) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]

23. Primary Outcome: Main Study: Percentage of Responders for Envelope (Env)-Specific Binding Antibody Titers at Week 72
Description: as for outcome 21
Time Frame: Week 72
Population: PPI set was used. Here, "N" (Number of participants analyzed): participants evaluable for this outcome measure and 'n' (number analyzed): number of participants analyzed for specified categories.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 16 | 77 | 18
percentage of responders
  Clade B (SC42261): number analyzed (Participants) | 16 | 76 | 18
  Clade B (SC42261) | 93.8 [69.8 to 99.8] | 94.7 [87.1 to 98.5] | 0 [0 to 0]
  Clade C (CH505TF): number analyzed (Participants) | 16 | 76 | 18
  Clade C (CH505TF) | 100 [78.2 to 100] | 96.1 [89 to 99.2] | 0 [0 to 0]
  Clade A (9004S): number analyzed (Participants) | 15 | 77 | 18
  Clade A (9004S) | 100 [78.2 to 100] | 100 [95.2 to 100] | 0 [0 to 0]
  Clade B (RHPA): number analyzed (Participants) | 15 | 77 | 18
  Clade B (RHPA) | 100 [78.2 to 100] | 100 [95.3 to 100] | 0 [0 to 0]
  Clade B (WITO): number analyzed (Participants) | 15 | 77 | 18
  Clade B (WITO) | 100 [78.2 to 100] | 100 [95.3 to 100] | 0 [0 to 0]
  Clade C (1086C): number analyzed (Participants) | 15 | 77 | 18
  Clade C (1086C) | 100 [78.2 to 100.0] | 100 [95.3 to 100.0] | 0 [0 to 0]
  Clade C (BF1266): number analyzed (Participants) | 15 | 77 | 18
  Clade C (BF1266) | 100 [78.2 to 100.0] | 98.7 [93 to 100.0] | 0 [0 to 0]
  CladeAE (conAE): number analyzed (Participants) | 15 | 77 | 18
  CladeAE (conAE) | 100 [78.2 to 100] | 97.4 [90.9 to 99.7] | 0 [0 to 0]
  Clade M(Con S): number analyzed (Participants) | 15 | 77 | 18
  Clade M(Con S) | 100 [78.2 to 100] | 100 [95.3 to 100] | 0 [0 to 0]

24. Primary Outcome: Late-boost (LB) Vaccination Phase: Geometric Mean of Envelope (Env) Mos 1 Specific Binding Antibodies (Abs) Response as Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 192
Description: Geometric mean of Env Mos 1 specific binding Abs response at Week 192 were assessed using ELISA.
Time Frame: Week 192
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit). Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Groups:
- Group 1b:LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study): Participants from Group 1 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with Ad26.Mos4.HIV and bivalent gp140 containing adjuvanted protein co-formulation with 80 mcg Clade C protein, 75 mcg Mosaic protein and 425 mcg aluminum (as aluminum phosphate adjuvant) as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
- Group 2b: LTE Then LB: Placebo (Previously in Group 1 of Main Study): Participants from Group 1 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with placebo matching to Ad26.Mos4.HIV and matching to gp140 HIV bivalent as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
- Group 1b:LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study): Participants from Group 2 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with Ad26.Mos4.HIV and bivalent gp140 containing adjuvanted protein co-formulation with 80 mcg Clade C protein, 75 mcg Mosaic protein and 425 mcg aluminum (as aluminum phosphate adjuvant) as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
- Group 2b: LTE Then LB: Placebo (Previously in Group 2 of Main Study): Participants from Group 1 and 2 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with placebo matching to Ad26.Mos4.HIV and matching to gp140 HIV bivalent as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
Arm/Group | Group 1b:LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 1 of Main Study) | Group 1b:LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 2 of Main Study)
Number analyzed (Participants) | 8 | 3 | 33 | 9
ELISA units/milliliter (EU/mL) | 4044.7 [2132.9 to 7670.2] | 3398.9 [979.0 to 11800.9] | 6816.4 [5125.4 to 9065.2] | 5125.0 [3079.4 to 8529.3]

25. Primary Outcome: Late-boost (LB) Vaccination Phase: Geometric Mean of Envelope (Env) Mos 1 Specific Binding Antibodies (Abs) Response as Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 193
Description: Geometric Mean of Env Mos 1 specific binding Abs response at Week 193 were assessed using ELISA.
Time Frame: Week 193
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Arm/Group | Group 1b:LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 1 of Main Study) | Group 1b:LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 2 of Main Study)
Number analyzed (Participants) | 8 | 2 | 32 | 9
ELISA units/milliliter (EU/mL) | 28412.2 [7194.6 to 112202.7] | 3652.9 [7.7 to 1726909.7] | 46851.6 [26104.6 to 84087.6] | 4505.3 [3439.9 to 5900.6]

26. Primary Outcome: Late-boost (LB) Vaccination Phase: Geometric Mean of Envelope (Env) Mos 1 Specific Binding Antibodies (Abs) Response as Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 196
Description: Geometric mean of Env Mos 1 specific binding Abs response at Week 196 were assessed using ELISA.
Time Frame: Week 196
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Groups:
- Group 1b: LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study): Participants from Group 1 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with Ad26.Mos4.HIV and bivalent gp140 containing adjuvanted protein co-formulation with 80 mcg Clade C protein, 75 mcg Mosaic protein and 425 mcg aluminum (as aluminum phosphate adjuvant) as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
- Group 1b: LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study): Participants from Group 2 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with Ad26.Mos4.HIV and bivalent gp140 containing adjuvanted protein co-formulation with 80 mcg Clade C protein, 75 mcg Mosaic protein and 425 mcg aluminum (as aluminum phosphate adjuvant) as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
Arm/Group | Group 1b: LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 1 of Main Study) | Group 1b: LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 2 of Main Study)
Number analyzed (Participants) | 7 | 3 | 32 | 10
ELISA units/milliliter (EU/mL) | 169017.3 [102848.8 to 277755.8] | 3438.1 [1190.8 to 9926.6] | 174004.6 [124094.4 to 243988.4] | 5153.9 [3377.6 to 7864.4]

27. Primary Outcome: Late-boost (LB) Vaccination Phase: Geometric Mean of Envelope (Env) Mos 1 Specific Binding Antibodies (Abs) Response as Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 204
Description: Geometric mean of Env Mos 1 specific binding Abs response at Week 204 were assessed using ELISA.
Time Frame: Week 204
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Groups:
- Group 1b:LTE Then LB: Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study): Participants from Group 1 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with Ad26.Mos4.HIV and bivalent gp140 containing adjuvanted protein co-formulation with 80 mcg Clade C protein, 75 mcg Mosaic protein and 425 mcg aluminum (as aluminum phosphate adjuvant) as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
- Group 1b:LTE Then LB: Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study): Participants from Group 2 of main study that entered the LTE phase were offered to enter in extension of LTE phase (late boost vaccination phase) and received late- boost vaccination with Ad26.Mos4.HIV and bivalent gp140 containing adjuvanted protein co-formulation with 80 mcg Clade C protein, 75 mcg Mosaic protein and 425 mcg aluminum (as aluminum phosphate adjuvant) as IM injection within 4 weeks prior to Week 192 until 4 months after Week 192 (that is, any day from Week 188 to Week 208) and were followed up until Week 288.
Arm/Group | Group 1b:LTE Then LB: Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 1 of Main Study) | Group 1b:LTE Then LB: Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 2 of Main Study)
Number analyzed (Participants) | 8 | 3 | 31 | 10
ELISA units/milliliter (EU/mL) | 65259.8 [35974.8 to 118383.9] | 3440.8 [835.5 to 14170.2] | 74715.2 [51288.6 to 108842.1] | 5303.2 [3435.7 to 8185.7]

28. Primary Outcome: Late-boost (LB) Vaccination Phase: Geometric Mean of Envelope (Env) Mos 1 Specific Binding Antibodies (Abs) Response as Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 216
Description: Geometric mean of Env Mos 1 specific binding Abs response at Week 216 were assessed using ELISA.
Time Frame: Week 216
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Arm/Group | Group 1b:LTE Then LB: Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 1 of Main Study) | Group 1b: LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 2 of Main Study)
Number analyzed (Participants) | 8 | 2 | 33 | 9
ELISA units/milliliter (EU/mL) | 27307.4 [12695.8 to 58735.4] | 3237.3 [4.2 to 2511983.7] | 43831.8 [30033.5 to 63969.3] | 5029.6 [3219.4 to 7857.7]

29. Primary Outcome: Late-boost (LB) Vaccination Phase: Geometric Mean of Envelope (Env) Mos 1 Specific Binding Antibodies (Abs) Response as Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 240
Description: Geometric mean of Env Mos 1 specific binding Abs response at Week 240 were assessed using ELISA.
Time Frame: Week 240
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Arm/Group | Group 1b: LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 1 of Main Study) | Group 1b:LTE Then LB: Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 2 of Main Study)
Number analyzed (Participants) | 8 | 2 | 33 | 9
ELISA units/milliliter (EU/mL) | 18223.4 [8647.7 to 38402.3] | 3031.1 [19.6 to 467682.9] | 25693.2 [17757.9 to 37174.7] | 4491.1 [2492.1 to 8093.7]

30. Primary Outcome: Late-boost (LB) Vaccination Phase: Geometric Mean of Envelope (Env) Mos 1 Specific Binding Antibodies (Abs) Response as Assessed Using Enzyme-linked Immunosorbent Assay (ELISA) at Week 288
Description: Geometric mean of Env Mos 1 specific binding Abs response at Week 288 were assessed using ELISA.
Time Frame: Week 288
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/milliliter (EU/mL)
Arm/Group | Group 1b: LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 1 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 1 of Main Study) | Group 1b: LTE Then LB:Ad26.Mos4.HIV+gp140 HIV Bivalent Vaccine (Previously in Group 2 of Main Study) | Group 2b: LTE Then LB: Placebo (Previously in Group 2 of Main Study)
Number analyzed (Participants) | 6 | 1 | 22 | 8
ELISA units/milliliter (EU/mL) | 18799.1 [8267.1 to 42748.8] | 4742.3 [NA to NA] — NA refers to lower and upper limits of 95% CI were not applicable for single participant. | 15757.0 [10438.7 to 23784.7] | 3933.1 [2772.2 to 5580.2]

31. Secondary Outcome: Main Study: Percentage of Responders of Env-Specific Neutralizing Antibody (nAbs) for Tier 1 Viruses
Description: Percentage of responders of Env-specific nAbs for tier 1 viruses were reported. Viruses with a Tier 1 neutralization phenotype: Clade C: MW965 and 97ZA012, ZM233M, CE703010010, 2759058, ZM215F, SO431, CE704810053 were used. The response was defined as post-baseline value >LLOQ.
Time Frame: Weeks 28, 52, and 72 (only for Clade C [MW965])
Population: PPI set was used in this analysis. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed for specified timepoints. n=0 signifies no participant was available for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Groups:
- Group 1: Ad26.Mos4.HIV + Clade C gp140: Participants received single intramuscular (IM) injection of Ad26.Mos4.HIV vaccine 5*10^10 viral particles (vp) at Weeks 0 and 12, followed by Ad26.Mos4.HIV vaccine 5*10^10 vp + Clade C glycoprotein 140 vaccine containing 250 micrograms (mcg) of total protein mixed with adjuvant (aluminum phosphate) IM injection at Weeks 24 and 48. Participants who received all 4 vaccinations and were negative for HIV infection at Week 72 and consented separately for an optional long-term extension (LTE) phase after Week 72 and were followed up until Week 216 (for participants who did not enter late boost vaccination phase) and up to any day between Week 188 to Week 208 for those who entered late boost extension.
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 20 | 90 | 25
Percentage of responders
  Clade C (MW965): Week 28 | 100.0 [83.2 to 100.0] | 100.0 [96.0 to 100.0] | 0 [0 to 0]
  Clade C (MW965): Week 52: number analyzed (Participants) | 17 | 81 | 23
  Clade C (MW965): Week 52 | 100.0 [80.5 to 100.0] | 100.0 [95.5 to 100.0] | 0 [0 to 0]
  Clade C (MW965) Week 72: number analyzed (Participants) | 17 | 79 | 0
  Clade C (MW965) Week 72 | 100.0 [80.5 to 100.0] | 98.7 [93.1 to 100.0] |
  Clade C (97ZA012): Week 28 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Clade C (97ZA012): Week 52: number analyzed (Participants) | 17 | 81 | 23
  Clade C (97ZA012): Week 52 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Clade C (ZM233M): Week 28: number analyzed (Participants) | 4 | 10 | 0
  Clade C (ZM233M): Week 28 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (ZM233M): Week 52: number analyzed (Participants) | 4 | 18 | 0
  Clade C (ZM233M): Week 52 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (CE703010010): Week 28: number analyzed (Participants) | 4 | 10 | 0
  Clade C (CE703010010): Week 28 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (CE703010010): Week 52: number analyzed (Participants) | 4 | 18 | 0
  Clade C (CE703010010): Week 52 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (2759058): Week 28: number analyzed (Participants) | 4 | 10 | 0
  Clade C (2759058): Week 28 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (2759058): Week 52: number analyzed (Participants) | 4 | 18 | 0
  Clade C (2759058): Week 52 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (ZM215F): Week 28: number analyzed (Participants) | 4 | 10 | 0
  Clade C (ZM215F): Week 28 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (ZM215F): Week 52: number analyzed (Participants) | 4 | 18 | 0
  Clade C (ZM215F): Week 52 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (SO431): Week 28: number analyzed (Participants) | 4 | 10 | 0
  Clade C (SO431): Week 28 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (SO431): Week 52: number analyzed (Participants) | 4 | 18 | 0
  Clade C (SO431): Week 52 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C (CE704810053): Week 28: number analyzed (Participants) | 4 | 10 | 0
  Clade C (CE704810053): Week 28 | 0 [0 to 0] | 0 [0 to 0] |
  Clade C(CE704810053): Week 52: number analyzed (Participants) | 4 | 18 | 0
  Clade C(CE704810053): Week 52 | 0 [0 to 0] | 0 [0 to 0] |

32. Secondary Outcome: Long-term Extension (LTE) Phase: Percentage of Responders of Env-Specific Neutralizing Antibody (nAbs) for Tier 1 Viruses
Description: Percentage of responders of Env-specific nAbs for tier 1 viruses were planned to be reported.
Time Frame: From Week 72 to Week 216
Population: LTE analysis set included all participants in the PPI Analysis set who were enrolled in the LTE phase of the study. Participants who received the late-boost vaccination were excluded from Week 192 onwards. Per change in planned analysis, data was not collected and analyzed due to limited scientific merit in the interpretation of this outcome measure.
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Late-boost (LB) Vaccination Phase: Percentage of Responders of Env-Specific Neutralizing Antibody (nAbs) for Tier 1 Viruses
Description: Percentage of responders of Env-specific nAbs for tier 1 viruses were planned to be reported.
Time Frame: From Week 188 up to end of study (Week 288)
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit). Per change in planned analysis, data was not collected and analyzed due to limited scientific merit in the interpretation of this outcome measure.
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Main Study: Percentage of Responders for Env-Specific Functional Antibody Response (Env ADCP gp140)
Description: Percentage of responders for Env-specific functional antibody response (Env ADCP gp140) were reported. The response was defined as post-baseline value > limit of detection (LOD) if baseline value <LOD or missing or defined as post-baseline value >3-fold increase from baseline if baseline value >=LOD. The lower limits of detection (LODs) for this assay were 5.16, 6.43, 6.49, 4.32 and 4.28 (phagocytic score) for Clade A (92UG037.1), Clade B (1990a), Clade C (Con C), Clade C (ZA), and Mos1, respectively.
Time Frame: Weeks 28, 52, and 72 (Weeks 52 and 72 are only for HIV ENV [gp140 T sortA] C [ZA] F Ab)
Population: PPI set was used in this analysis. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed for specified timepoints.
Measure: Number; unit: Percentage of Responders
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 23 | 92 | 25
Percentage of Responders
  HIV ENV (gp140 M sortA) A (92UG037) F Ab: Week 28: number analyzed (Participants) | 20 | 90 | 25
  HIV ENV (gp140 M sortA) A (92UG037) F Ab: Week 28 | 90.0 | 94.4 | 32.0
  HIV ENV (gp140 M sortA) B (1990a) F Ab: Week 28: number analyzed (Participants) | 20 | 90 | 25
  HIV ENV (gp140 M sortA) B (1990a) F Ab: Week 28 | 90.0 | 98.9 | 0
  HIV ENV (gp140 M sortA) C (conC) F Ab: Week 28: number analyzed (Participants) | 20 | 90 | 25
  HIV ENV (gp140 M sortA) C (conC) F Ab: Week 28 | 85.0 | 91.1 | 0
  HIV ENV (gp140 T sortA) (Mos1) F Ab: Week 28: number analyzed (Participants) | 20 | 90 | 25
  HIV ENV (gp140 T sortA) (Mos1) F Ab: Week 28 | 100.0 | 100.0 | 36.0
  HIV ENV (gp140 T sortA) C (ZA) F Ab: Week 28 | 95.0 | 100.0 | 8.0
  HIV ENV (gp140 T sortA) C (ZA) F Ab: Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV ENV (gp140 T sortA) C (ZA) F Ab: Week 52 | 100.0 | 100.0 | 13.0
  HIV ENV (gp140 T sortA) C (ZA) F Ab: Week 72: number analyzed (Participants) | 17 | 84 | 21
  HIV ENV (gp140 T sortA) C (ZA) F Ab: Week 72 | 100.0 | 96.4 | 52.4

35. Secondary Outcome: Long-term Extension (LTE) Phase: Percentage of Responders for Env-Specific Functional Antibody Response (Env ADCP gp140)
Description: Percentage of responders for Env-specific functional antibody response (Env ADCP gp140) were planned to be reported.
Time Frame: From Week 72 up to Week 216
Population: as for outcome 32
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Late-boost (LB) Vaccination Phase: Percentage of Responders for Env-Specific Functional Antibody Response (Env ADCP gp140)
Description: Percentage of responders for Env-specific functional antibody response (Env ADCP gp140) were planned to be reported.
Time Frame: From Week 188 up to end of study (Week 288)
Population: as for outcome 33
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Main Study: Percentage of Responders for Env-Specific Binding Ab Isotypes (Immunoglobulin [Ig] G1 and IgG3)
Description: Percentage of responders for Env-specific binding Ab isotypes (IgG1 and IgG3) for Clade C (ZA) as assessed using ELISA were reported. The response was defined as post-baseline value >LLOQ if baseline <LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=LLOQ. The LLOQs for this assay were 12.3 and 12.4 EC50 for IgG1 and IgG3, respectively. EC50= 50% effective concentration.
Time Frame: Weeks 28, 52, and 72
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 20 | 90 | 25
Percentage of Responders
  HIV ENV (gp140 T) clade C (ZA) IgG-1 Ab: Week 28 | 65.0 [40.8 to 84.6] | 76.7 [66.6 to 84.9] | 0 [0 to 0]
  HIV ENV (gp140 T) clade C (ZA) IgG-1 Ab: Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV ENV (gp140 T) clade C (ZA) IgG-1 Ab: Week 52 | 76.5 [50.1 to 93.2] | 75.6 [64.9 to 84.4] | 0 [0 to 0]
  HIV ENV (gp140 T) clade C (ZA) IgG-1 Ab: Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV ENV (gp140 T) clade C (ZA) IgG-1 Ab: Week 72 | 76.5 [50.1 to 93.2] | 66.3 [55.1 to 76.3] | 0 [0 to 0]
  HIV ENV (gp140 T) clade C (ZA) IgG-3 Ab: Week 28: number analyzed (Participants) | 20 | 88 | 23
  HIV ENV (gp140 T) clade C (ZA) IgG-3 Ab: Week 28 | 60.0 [36.1 to 80.9] | 75.0 [64.6 to 83.6] | 8.7 [1.1 to 28.0]
  HIV ENV (gp140 T) clade C (ZA) IgG-3 Ab: Week 52: number analyzed (Participants) | 16 | 82 | 23
  HIV ENV (gp140 T) clade C (ZA) IgG-3 Ab: Week 52 | 75.0 [47.6 to 92.7] | 73.2 [62.2 to 82.4] | 0 [0 to 0]
  HIV ENV (gp140 T) clade C (ZA) IgG-3 Ab: Week 72: number analyzed (Participants) | 17 | 82 | 21
  HIV ENV (gp140 T) clade C (ZA) IgG-3 Ab: Week 72 | 23.5 [6.8 to 49.9] | 36.6 [26.2 to 48.0] | 14.3 [3.0 to 36.3]

38. Secondary Outcome: Long-term Extension (LTE) Phase: Percentage of Responders for Env-Specific Binding Ab Isotypes (Immunoglobulin [Ig] G1 and IgG3)
Description: Percentage of responders for Env-specific binding Ab isotypes IgG1 and IgG3) were planned to be reported.
Time Frame: From Week 72 up to Week 216
Population: as for outcome 32
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Late-boost (LB) Vaccination Phase: Percentage of Responders for Env-Specific Binding Ab Isotypes (Immunoglobulin [Ig] G1 and IgG3)
Description: Percentage of responders for Env-specific binding Ab isotypes IgG1 and IgG3) were planned to be reported.
Time Frame: From Week 188 up to end of study (Week 288)
Population: as for outcome 33
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Main Study: Percentage of Interferon (IFN)-Gamma Peripheral Blood Mononuclear Cell (PBMC) Responders to Mosaic and Potential T-cell Epitope (PTE) Peptide Pools of Env/Group-Specific Antigen (Gag)/ Polymerase (Pol)
Description: Percentage of IFN-gamma PBMC responders to mosaic and PTE peptide pools of Env/Gag/Pol as assessed by ELISpot was reported. The response was defined as post-baseline value >P95 if baseline <P95 or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=P95.
Time Frame: Weeks 28, 52, and 72
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 21 | 89 | 25
Percentage of Responders
  HIV IFNg ENV pep pool (Clinical PTE): Week 28 | 90.5 [69.6 to 98.8] | 82.0 [72.5 to 89.4] | 0 [0 to 0]
  HIV IFNg ENV pep pool (Clinical PTE): Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV IFNg ENV pep pool (Clinical PTE): Week 52 | 82.4 [56.6 to 96.2] | 87.8 [78.7 to 94.0] | 4.3 [0.1 to 21.9]
  HIV IFNg ENV pep pool (Clinical PTE): Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV IFNg ENV pep pool (Clinical PTE): Week 72 | 76.5 [50.1 to 93.2] | 84.3 [74.7 to 91.4] | 4.8 [0.1 to 23.8]
  HIV IFNg ENV pep pool (Mos1): Week 28 | 90.5 [69.6 to 98.8] | 85.4 [76.3 to 92.0] | 4.0 [0.1 to 20.4]
  HIV IFNg ENV pep pool (Mos1): Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV IFNg ENV pep pool (Mos1): Week 52 | 94.1 [71.3 to 99.9] | 84.1 [74.4 to 91.3] | 13.0 [2.8 to 33.6]
  HIV IFNg ENV pep pool (Mos1): Week 72: number analyzed (Participants) | 14 | 78 | 20
  HIV IFNg ENV pep pool (Mos1): Week 72 | 85.7 [57.2 to 98.2] | 85.9 [76.2 to 92.7] | 10.0 [1.2 to 31.7]
  HIV IFNg ENV pep pool (Mos2): Week 28 | 81.0 [58.1 to 94.6] | 88.8 [80.3 to 94.5] | 4.0 [0.1 to 20.4]
  HIV IFNg ENV pep pool (Mos2): Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV IFNg ENV pep pool (Mos2): Week 52 | 94.1 [71.3 to 99.9] | 87.8 [78.7 to 94.0] | 8.7 [1.1 to 28.0]
  HIV IFNg ENV pep pool (Mos2): Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV IFNg ENV pep pool (Mos2): Week 72 | 70.6 [44.0 to 89.7] | 86.7 [77.5 to 93.2] | 4.8 [0.1 to 23.8]
  HIV IFNg Gag pep pool (Clinical PTE) : Week 28 | 52.4 [29.8 to 74.3] | 31.5 [22.0 to 42.2] | 0 [0 to 0]
  HIV IFNg Gag pep pool (Clinical PTE) : Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV IFNg Gag pep pool (Clinical PTE) : Week 52 | 41.2 [18.4 to 67.1] | 32.9 [22.9 to 44.2] | 0 [0 to 0]
  HIV IFNg Gag pep pool (Clinical PTE) : Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV IFNg Gag pep pool (Clinical PTE) : Week 72 | 41.2 [18.4 to 67.1] | 26.5 [17.4 to 37.3] | 0 [0 to 0]
  HIV IFNg Gag pep pool (Mos1): Week 28 | 52.4 [29.8 to 74.3] | 56.2 [45.3 to 66.7] | 4.0 [0.1 to 20.4]
  HIV IFNg Gag pep pool (Mos1): Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV IFNg Gag pep pool (Mos1): Week 52 | 52.9 [27.8 to 77.0] | 51.2 [39.9 to 62.4] | 4.3 [0.1 to 21.9]
  HIV IFNg Gag pep pool (Mos1): Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV IFNg Gag pep pool (Mos1): Week 72 | 52.9 [27.8 to 77.0] | 48.2 [37.1 to 59.4] | 4.8 [0.1 to 23.8]
  HIV IFNg Gag pep pool (Mos2): Week 28 | 61.9 [38.4 to 81.9] | 60.7 [49.7 to 70.9] | 8.0 [1.0 to 26.0]
  HIV IFNg Gag pep pool (Mos2): Week 52: number analyzed (Participants) | 16 | 82 | 23
  HIV IFNg Gag pep pool (Mos2): Week 52 | 75.0 [47.6 to 92.7] | 52.4 [41.1 to 63.6] | 8.7 [1.1 to 28.0]
  HIV IFNg Gag pep pool (Mos2): Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV IFNg Gag pep pool (Mos2): Week 72 | 58.8 [32.9 to 81.6] | 47.0 [35.9 to 58.3] | 0 [0 to 0]
  HIV IFNg Pol pep pool (Clinical PTE): Week 28 | 76.2 [52.8 to 91.8] | 77.5 [67.4 to 85.7] | 4.0 [0.1 to 20.4]
  HIV IFNg Pol pep pool (Clinical PTE): Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV IFNg Pol pep pool (Clinical PTE): Week 52 | 82.4 [56.6 to 96.2] | 86.6 [77.3 to 93.1] | 4.3 [0.1 to 21.9]
  HIV IFNg Pol pep pool (Clinical PTE): Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV IFNg Pol pep pool (Clinical PTE): Week 72 | 76.5 [50.1 to 93.2] | 83.1 [73.3 to 90.5] | 0 [0 to 0]
  HIV IFNg Pol pep pool (Mos1): Week 28 | 76.2 [52.8 to 91.8] | 75.3 [65.0 to 83.8] | 8.0 [1.0 to 26.0]
  HIV IFNg Pol pep pool (Mos1): Week 52: number analyzed (Participants) | 17 | 82 | 23
  HIV IFNg Pol pep pool (Mos1): Week 52 | 58.8 [32.9 to 81.6] | 78.0 [67.5 to 86.4] | 17.4 [5.0 to 38.8]
  HIV IFNg Pol pep pool (Mos1): Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV IFNg Pol pep pool (Mos1): Week 72 | 47.1 [23.0 to 72.2] | 73.5 [62.7 to 82.6] | 0 [0 to 0]
  HIV IFNg Pol pep pool (Mos2): Week 28 | 76.2 [52.8 to 91.8] | 83.1 [73.7 to 90.2] | 4.0 [0.1 to 20.4]
  HIV IFNg Pol pep pool (Mos2): Week 52: number analyzed (Participants) | 16 | 82 | 23
  HIV IFNg Pol pep pool (Mos2): Week 52 | 75.0 [47.6 to 92.7] | 85.4 [75.8 to 92.2] | 17.4 [5.0 to 38.8]
  HIV IFNg Pol pep pool (Mos2): Week 72: number analyzed (Participants) | 17 | 83 | 21
  HIV IFNg Pol pep pool (Mos2): Week 72 | 70.6 [44.0 to 89.7] | 80.7 [70.6 to 88.6] | 9.5 [1.2 to 30.4]

41. Secondary Outcome: Long-term Extension (LTE) Phase: Percentage of Interferon (IFN)-Gamma Peripheral Blood Mononuclear Cell (PBMC) Responders to Mosaic and Potential T-cell Epitope (PTE) Peptide Pools of Env/Group-Specific Antigen (Gag)/ Polymerase (Pol)
Description: Percentage of Interferon (IFN)-Gamma PBMC responders to Mosaic and Potential T-cell Epitope (PTE) Peptide Pools of Env/Group-Specific Antigen (Gag)/ Polymerase (Pol) was planned to be reported.
Time Frame: From Week 72 up to Week 216
Population: as for outcome 32
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Late-boost (LB) Vaccination Phase: Percentage of Interferon (IFN)-Gamma Peripheral Blood Mononuclear Cell (PBMC) Responders to Mosaic and Potential T-cell Epitope (PTE) Peptide Pools of Env/Group-Specific Antigen (Gag)/ Polymerase (Pol)
Description: Percentage of Interferon (IFN)-Gamma PBMC responders to Mosaic and Potential T-cell Epitope (PTE) Peptide Pools of Env/Group-Specific Antigen (Gag)/ Polymerase (Pol) were planned to be reported.
Time Frame: From Week 188 up to end of study (Week 288)
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit) was planned to be used. Per change in planned analysis, data was not collected and analyzed due to limited scientific merit in the interpretation of this outcome measure.
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Main Study: Percentage of Responders With Cluster of Differentiation (CD)4+ and CD8+ T-Cell Functionality
Description: Percentage of responders with CD4+ and CD8+ T-cell functionality (cells producing IFN-gamma and /or IL-2) were reported. Intracellular cytokine staining (ICS) was performed to examine the type of T-cell responding to vaccination. Responder definition was based on the Fisher's exact text between cytokine producing cells and non-producing cells in stimulated versus non-stimulated conditions.
Time Frame: Weeks 28, 52, and 72
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3: Placebo
Number analyzed (Participants) | 20 | 87 | 24
Percentage of responders
  CD4+: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4+: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 28 | 50.00 [27.20 to 72.80] | 80.95 [70.92 to 88.70] | 0 [0 to 0]
  CD4+: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4+: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 52 | 64.29 [35.14 to 87.24] | 77.46 [66.00 to 86.54] | 0 [0 to 0]
  CD4+: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4+: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 72 | 41.18 [18.44 to 67.08] | 69.23 [57.76 to 79.19] | 0 [0 to 0]
  CD4+: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4+: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 28 | 50.00 [27.20 to 72.80] | 80.95 [70.92 to 88.70] | 0 [0 to 0]
  CD4+: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4+: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 52 | 64.29 [35.14 to 87.24] | 74.65 [62.92 to 84.23] | 0 [0 to 0]
  CD4+: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4+: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 72 | 29.41 [10.31 to 55.96] | 69.23 [57.76 to 79.19] | 0 [0 to 0]
  CD4+: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4+: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28 | 40.00 [19.12 to 63.95] | 53.57 [42.35 to 64.53] | 0 [0 to 0]
  CD4+: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4+: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52 | 57.14 [28.86 to 82.34] | 47.89 [35.88 to 60.08] | 0 [0 to 0]
  CD4+: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4+: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72 | 29.41 [10.31 to 55.96] | 21.79 [13.24 to 32.59] | 0 [0 to 0]
  CD4+: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4+: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 28 | 50.00 [27.20 to 72.80] | 82.14 [72.26 to 89.65] | 0 [0 to 0]
  CD4+: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4+: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 52 | 64.29 [35.14 to 87.24] | 77.46 [66.00 to 86.54] | 0 [0 to 0]
  CD4+: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4+: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 72 | 41.18 [18.44 to 67.08] | 69.23 [57.76 to 79.19] | 0 [0 to 0]
  CD4+: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4+: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 28 | 10.00 [1.23 to 31.70] | 8.33 [3.42 to 16.42] | 0 [0 to 0]
  CD4+: HIV Gag pep pool ANY: Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4+: HIV Gag pep pool ANY: Week 52 | 7.14 [0.18 to 33.87] | 9.86 [4.06 to 19.26] | 0 [0 to 0]
  CD4+: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4+: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 72 | 5.88 [0.15 to 28.69] | 1.28 [0.03 to 6.94] | 0 [0 to 0]
  CD4+: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4+: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 28 | 10.00 [1.23 to 31.70] | 8.33 [3.42 to 16.42] | 0 [0 to 0]
  CD4+: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4+: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 52 | 0 [0 to 0] | 11.27 [4.99 to 21.00] | 0 [0 to 0]
  CD4+: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4+: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 72 | 0 [0 to 0] | 1.28 [0.03 to 6.94] | 0 [0 to 0]
  CD4 +: HIV ENV gp120 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4 +: HIV ENV gp120 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28 | 50.00 [27.20 to 72.80] | 80.95 [70.92 to 88.70] | 0 [0 to 0]
  CD4 +: HIV ENV gp120 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4 +: HIV ENV gp120 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52 | 57.14 [28.86 to 82.34] | 73.24 [61.41 to 83.06] | 0 [0 to 0]
  CD4 +: HIV ENV gp120 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4 +: HIV ENV gp120 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72 | 29.41 [10.31 to 55.96] | 69.23 [57.76 to 79.19] | 0 [0 to 0]
  CD4 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28 | 40.00 [19.12 to 63.95] | 47.62 [36.60 to 58.81] | 0 [0 to 0]
  CD4 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52 | 42.86 [17.66 to 71.14] | 43.66 [31.91 to 55.95] | 0 [0 to 0]
  CD4 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72 | 23.53 [6.81 to 49.90] | 19.23 [11.18 to 29.73] | 0 [0 to 0]
  CD4 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 82 | 23
  CD4 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28 | 15.79 [3.38 to 39.58] | 28.05 [18.68 to 39.06] | 0 [0 to 0]
  CD4 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52 | 21.43 [4.66 to 50.80] | 19.72 [11.22 to 30.86] | 0 [0 to 0]
  CD4 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72 | 5.88 [0.15 to 28.69] | 12.82 [6.32 to 22.32] | 0 [0 to 0]
  CD4 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28 | 20.00 [5.73 to 43.66] | 32.14 [22.36 to 43.22] | 0 [0 to 0]
  CD4 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52 | 42.86 [17.66 to 71.14] | 23.94 [14.61 to 35.54] | 0 [0 to 0]
  CD4 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72 | 5.88 [0.15 to 28.69] | 10.26 [4.53 to 19.21] | 0 [0 to 0]
  CD4 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 28 | 10.00 [1.23 to 31.70] | 8.33 [3.42 to 16.42] | 0 [0 to 0]
  CD4 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 52 | 7.14 [0.18 to 33.87] | 9.86 [4.06 to 19.26] | 0 [0 to 0]
  CD4 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 72 | 5.88 [0.15 to 28.69] | 1.28 [0.03 to 6.94] | 0 [0 to 0]
  CD4 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28 | 10.00 [1.23 to 31.70] | 2.38 [0.29 to 8.34] | 0 [0 to 0]
  CD4 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52 | 0 [0 to 0] | 7.04 [2.33 to 15.67] | 0 [0 to 0]
  CD4 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72 | 0 [0 to 0] | 1.28 [0.03 to 6.94] | 0 [0 to 0]
  CD4 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 20 | 84 | 24
  CD4 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 28 | 10.00 [1.23 to 31.70] | 5.95 [1.96 to 13.35] | 0 [0 to 0]
  CD4 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 14 | 71 | 21
  CD4 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 52 | 0 [0 to 0] | 7.04 [2.33 to 15.67] | 0 [0 to 0]
  CD4 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 78 | 19
  CD4 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 72 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  CD8 +: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 28 | 21.05 [6.05 to 45.57] | 33.33 [23.58 to 44.25] | 0 [0 to 0]
  CD8+: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8+: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 52 | 29.41 [10.31 to 55.96] | 29.11 [19.43 to 40.42] | 0 [0 to 0]
  CD8 +: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +: HIV ENV pep pool (Mos1 ZA) IFNg+ or IL2+ (%): Week 72 | 17.65 [3.80 to 43.43] | 26.25 [17.04 to 37.29] | 0 [0 to 0]
  CD8 +: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 28 | 10.53 [1.30 to 33.14] | 29.89 [20.54 to 40.65] | 0 [0 to 0]
  CD8 +: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 52 | 11.76 [1.46 to 36.44] | 26.58 [17.27 to 37.72] | 0 [0 to 0]
  CD8+: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8+: HIV ENV pep pool (Mos1) IFNg+ or IL2+ (%): Week 72 | 5.88 [0.15 to 28.69] | 25.00 [15.99 to 35.94] | 0 [0 to 0]
  CD8 +: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28 | 15.79 [3.38 to 39.58] | 14.94 [8.20 to 24.20] | 0 [0 to 0]
  CD8 +: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52 | 29.41 [10.31 to 55.96] | 13.92 [7.16 to 23.55] | 0 [0 to 0]
  CD8 +: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +: HIV ENV pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72 | 17.65 [3.80 to 43.43] | 13.75 [7.07 to 23.27] | 0 [0 to 0]
  CD8 +: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 28 | 73.68 [48.80 to 90.85] | 58.62 [47.55 to 69.08] | 0 [0 to 0]
  CD8 +: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 52 | 70.59 [44.04 to 89.69] | 58.23 [46.59 to 69.23] | 0 [0 to 0]
  CD8 +: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +: HIV Env Pol Gag pep pool IFNg+ or IL2+ (%): Week 72 | 52.94 [27.81 to 77.02] | 52.50 [41.02 to 63.79] | 0 [0 to 0]
  CD8 +: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 28 | 36.84 [16.29 to 61.64] | 21.84 [13.69 to 31.98] | 0 [0 to 0]
  CD8 +: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 52 | 35.29 [14.21 to 61.67] | 22.78 [14.10 to 33.60] | 0 [0 to 0]
  CD8 +: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +: HIV Gag pep pool ANY IFNg+ or IL2+ (%): Week 72 | 29.41 [10.31 to 55.96] | 17.50 [9.91 to 27.62] | 0 [0 to 0]
  CD8 +: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 28 | 63.16 [38.36 to 83.71] | 47.13 [36.33 to 58.13] | 0 [0 to 0]
  CD8 +: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 52 | 58.82 [32.92 to 81.56] | 49.37 [37.92 to 60.86] | 0 [0 to 0]
  CD8 +: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +: HIV Pol pep pool (Mos1) IFNg+ or IL2+ (%): Week 72 | 29.41 [10.31 to 55.96] | 40.00 [29.20 to 51.56] | 0 [0 to 0]
  CD8 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28 | 15.79 [3.38 to 39.58] | 9.20 [4.05 to 17.32] | 0 [0 to 0]
  CD8 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52 | 29.41 [10.31 to 55.96] | 10.13 [4.47 to 18.98] | 0 [0 to 0]
  CD8 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +:HIV ENV gp120 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72 | 17.65 [3.80 to 43.43] | 8.75 [3.59 to 17.20] | 0 [0 to 0]
  CD8 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 18 | 85 | 23
  CD8 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28 | 5.56 [0.14 to 27.29] | 11.76 [5.79 to 20.57] | 0 [0 to 0]
  CD8 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52 | 0 [0 to 0] | 12.66 [6.24 to 22.05] | 0 [0 to 0]
  CD8 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +:HIV ENV gp41 pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72 | 0 [0 to 0] | 13.75 [7.07 to 23.27] | 0 [0 to 0]
  CD8 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 28 | 0 [0 to 0] | 9.20 [4.05 to 17.32] | 0 [0 to 0]
  CD8 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 52 | 0 [0 to 0] | 6.33 [2.09 to 14.16] | 0 [0 to 0]
  CD8 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +:HIV ENV gp41 pep pool clade C (ZA) IFNg+ or IL2+ (%): Week 72 | 0 [0 to 0] | 7.50 [2.80 to 15.61] | 0 [0 to 0]
  CD8 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 28 | 36.84 [16.29 to 61.64] | 21.84 [13.69 to 31.98] | 0 [0 to 0]
  CD8 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 52 | 35.29 [14.21 to 61.67] | 22.78 [14.10 to 33.60] | 0 [0 to 0]
  CD8 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +:HIV Gag pep pool (Mos1) IFNg+ or IL2+ (%): Week 72 | 29.41 [10.31 to 55.96] | 17.50 [9.91 to 27.62] | 0 [0 to 0]
  CD8 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 28 | 57.89 [33.50 to 79.75] | 29.89 [20.54 to 40.65] | 0 [0 to 0]
  CD8 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 52 | 47.06 [22.98 to 72.19] | 30.38 [20.53 to 41.75] | 0 [0 to 0]
  CD8 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +:HIV Pol RNAseInt pep pool 1 (Mos1) IFNg+ or IL2+ (%): Week 72 | 17.65 [3.80 to 43.43] | 20.00 [11.89 to 30.44] | 0 [0 to 0]
  CD8 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 28: number analyzed (Participants) | 19 | 87 | 24
  CD8 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 28 | 31.58 [12.58 to 56.55] | 31.03 [21.55 to 41.86] | 0 [0 to 0]
  CD8 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 52: number analyzed (Participants) | 17 | 79 | 23
  CD8 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 52 | 29.41 [10.31 to 55.96] | 30.38 [20.53 to 41.75] | 0 [0 to 0]
  CD8 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 72: number analyzed (Participants) | 17 | 80 | 20
  CD8 +:HIV Pol RT pep pool (Mos1) IFNg+ or IL2+ (%): Week 72 | 23.53 [6.81 to 49.90] | 27.50 [18.10 to 38.62] | 0 [0 to 0]

44. Secondary Outcome: Long-term Extension (LTE) Phase: Percentage of Responders With Cluster of Differentiation (CD)4+ and CD8+ T-Cell Functionality
Description: Percentage of Responders With Cluster of Differentiation (CD)4+ and CD8+ T-Cell Functionality (cells Producing IFN-Gamma and/or Interleukin [IL-2]) were planned to be reported. Intracellular cytokine staining (ICS) was performed to examine the type of T-cell responding to vaccination. Responder definition was based on the Fisher's exact text between cytokine producing cells and non-producing cells in stimulated versus non-stimulated conditions.
Time Frame: From Week 72 up to Week 216
Population: as for outcome 32
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Late-boost (LB) Vaccination Phase: Percentage of Responders With Cluster of Differentiation (CD)4+ and CD8+ T-Cell Functionality
Description: as for outcome 43
Time Frame: Weeks 192 and 196
Population: LB included all participants who received LB vaccination (at least one of the 2 vaccines at LB visit). Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed for specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 23 | 7
Percentage of responders
  CD4 +:Any Env IFNg+ or IL2+ (%): Week 192 | 82.6 [61.22 to 95.05] | 57.1 [18.41 to 90.10]
  CD4 +:Any Env IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:Any Env IFNg+ or IL2+ (%): Week 196 | 91.3 [71.96 to 98.93] | 83.3 [35.88 to 99.58]
  CD4 +:Any HIV IFNg+ or IL2+ (%): Week 192 | 82.6 [61.22 to 95.05] | 57.1 [18.41 to 90.10]
  CD4 +:Any HIV IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:Any HIV IFNg+ or IL2+ (%): Week 196 | 91.3 [71.96 to 98.93] | 83.3 [35.88 to 99.58]
  CD4 +:Any MOS1 Env IFNg+ or IL2+ (%): Week 192 | 73.9 [51.59 to 89.77] | 57.1 [18.41 to 90.10]
  CD4 +:Any MOS1 Env IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:Any MOS1 Env IFNg+ or IL2+ (%): Week 196 | 91.3 [71.96 to 98.93] | 83.3 [35.88 to 99.58]
  CD4 +:Any MOS2 Env IFNg+ or IL2+ (%): Week 192 | 65.2 [42.73 to 83.62] | 42.9 [9.90 to 81.59]
  CD4 +:Any MOS2 Env IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:Any MOS2 Env IFNg+ or IL2+ (%): Week 196 | 73.9 [51.59 to 89.77] | 33.3 [4.33 to 77.72]
  CD4 +:J Mos1 gp120 IFNg+ or IL2+ (%): Week 192 | 73.9 [51.59 to 89.77] | 57.1 [18.41 to 90.10]
  CD4 +:J Mos1 gp120 IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:J Mos1 gp120 IFNg+ or IL2+ (%): Week 196 | 91.3 [71.96 to 98.93] | 83.3 [35.88 to 99.58]
  CD4 +:J Mos1 gp41 IFNg+ or IL2+ (%): Week 192 | 39.1 [19.71 to 61.46] | 14.3 [0.36 to 57.87]
  CD4 +:J Mos1 gp41 IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:J Mos1 gp41 IFNg+ or IL2+ (%): Week 196 | 43.5 [23.19 to 65.51] | 33.3 [4.33 to 77.72]
  CD4 +:J Mos2 Gag IFNg+ or IL2+ (%): Week 192 | 21.7 [7.46 to 43.70] | 0 [0 to 0]
  CD4 +:J Mos2 Gag IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:J Mos2 Gag IFNg+ or IL2+ (%): Week 196 | 39.1 [19.71 to 61.46] | 0 [0 to 0]
  CD4 +:J Mos2 RNAseInt IFNg+ or IL2+ (%): Week 192 | 17.4 [4.95 to 38.78] | 0 [0 to 0]
  CD4 +:J Mos2 RNAseInt IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:J Mos2 RNAseInt IFNg+ or IL2+ (%): Week 196 | 17.4 [4.95 to 38.78] | 16.7 [0.42 to 64.12]
  CD4 +:J Mos2S gp120 IFNg+ or IL2+ (%): Week 192 | 60.9 [38.54 to 80.29] | 42.9 [9.90 to 81.59]
  CD4 +:J Mos2S gp120 IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:J Mos2S gp120 IFNg+ or IL2+ (%): Week 196 | 69.6 [47.08 to 86.79] | 33.3 [4.33 to 77.72]
  CD4 +:J Mos2S gp41 IFNg+ or IL2+ (%): Week 192 | 21.7 [7.46 to 43.70] | 0 [0 to 0]
  CD4 +:J Mos2S gp41 IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +:J Mos2S gp41 IFNg+ or IL2+ (%): Week 196 | 43.5 [23.19 to 65.51] | 16.7 [0.42 to 64.12]
  CD4 +: POSITIVE CONTROL (CMV) IFNg+ or IL2+ (%): Week 192 | 52.2 [30.59 to 73.18] | 57.1 [18.41 to 90.10]
  CD4 +: POSITIVE CONTROL (CMV) IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD4 +: POSITIVE CONTROL (CMV) IFNg+ or IL2+ (%): Week 196 | 50.0 [28.22 to 71.78] | 80.0 [28.36 to 99.49]
  CD8 +: Any HIV IFNg+ or IL2+ (%): Week 192 | 73.9 [51.59 to 89.77] | 28.6 [3.67 to 70.96]
  CD8 +: Any HIV IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: Any HIV IFNg+ or IL2+ (%): Week 196 | 73.9 [51.59 to 89.77] | 33.3 [4.33 to 77.72]
  CD8 +: Any MOS1 Env IFNg+ or IL2+ (%): Week 192 | 34.8 [16.38 to 57.27] | 14.3 [0.36 to 57.87]
  CD8 +: Any MOS1 Env IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: Any MOS1 Env IFNg+ or IL2+ (%): Week 196 | 43.5 [23.19 to 65.51] | 16.7 [0.42 to 64.12]
  CD8 +: Any MOS2 Env IFNg+ or IL2+ (%): Week 192 | 47.8 [26.82 to 69.41] | 14.3 [0.36 to 57.87]
  CD8 +: Any MOS2 Env IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: Any MOS2 Env IFNg+ or IL2+ (%): Week 196 | 47.8 [26.82 to 69.41] | 33.3 [4.33 to 77.72]
  CD8 +: J Mos1 gp120 IFNg+ or IL2+ (%): Week 192 | 17.4 [4.95 to 38.78] | 14.3 [0.36 to 57.87]
  CD8 +: J Mos1 gp120 IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: J Mos1 gp120 IFNg+ or IL2+ (%): Week 196 | 26.1 [10.23 to 48.41] | 16.7 [0.42 to 64.12]
  CD8 +: J Mos1 gp41 IFNg+ or IL2+ (%): Week 192 | 17.4 [4.95 to 38.78] | 0 [0 to 0]
  CD8 +: J Mos1 gp41 IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: J Mos1 gp41 IFNg+ or IL2+ (%): Week 196 | 21.7 [7.46 to 43.70] | 0 [0 to 0]
  CD8 +: J Mos2 Gag IFNg+ or IL2+ (%): Week 192 | 30.4 [13.21 to 52.92] | 0 [0 to 0]
  CD8 +: J Mos2 Gag IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: J Mos2 Gag IFNg+ or IL2+ (%): Week 196 | 30.4 [13.21 to 52.92] | 0 [0 to 0]
  CD8 +: J Mos2 RNAseInt IFNg+ or IL2+ (%): Week 192 | 34.8 [16.38 to 57.27] | 14.3 [0.36 to 57.87]
  CD8 +: J Mos2 RNAseInt IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: J Mos2 RNAseInt IFNg+ or IL2+ (%): Week 196 | 34.8 [16.38 to 57.27] | 16.7 [0.42 to 64.12]
  CD8 +: J Mos2S gp120 IFNg+ or IL2+ (%): Week 192 | 30.4 [13.21 to 52.92] | 14.3 [0.36 to 57.87]
  CD8 +: J Mos2S gp120 IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: J Mos2S gp120 IFNg+ or IL2+ (%): Week 196 | 34.8 [16.38 to 57.27] | 16.7 [0.42 to 64.12]
  CD8 +: J Mos2S gp41 IFNg+ or IL2+ (%): Week 192 | 17.4 [4.95 to 38.78] | 0 [0 to 0]
  CD8 +: J Mos2S gp41 IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 23 | 6
  CD8 +: J Mos2S gp41 IFNg+ or IL2+ (%): Week 196 | 17.4 [4.95 to 38.78] | 16.7 [0.42 to 64.12]
  CD8 +: POSITIVE CONTROL (CMV) IFNg+ or IL2+ (%): Week 192 | 52.2 [30.59 to 73.18] | 71.4 [29.04 to 96.33]
  CD8 +: POSITIVE CONTROL (CMV) IFNg+ or IL2+ (%): Week 196: number analyzed (Participants) | 22 | 5
  CD8 +: POSITIVE CONTROL (CMV) IFNg+ or IL2+ (%): Week 196 | 50.0 [28.22 to 71.78] | 80.0 [28.36 to 99.49]

46. Secondary Outcome: Main Study: Percentage of Participants With T-Cell Development
Description: Percentage of participants with T-Cell development were planned to be reported.
Time Frame: From Baseline (Day 1) up to Week 72
Population: PPI set included participants who received at least first 3 vaccines, as per protocol, had at least one measured post dose blood sample collected and were not diagnosed with HIV during study. Samples taken post Week 48 from participants in PPI set who missed or did not receive 4th vaccine in protocol specified time window (+/- 2 weeks) were excluded from analysis. Due to change in planned analysis, data was not collected and analyzed as assay was not qualified.
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Long-term Extension (LTE) Phase: Percentage of Participants With T-Cell Development
Description: Percentage of participants with T-Cell development were planned to be reported.
Time Frame: From Week 72 up to Week 216
Population: as for outcome 32
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C gp140 | Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Late-boost (LB) Vaccination Phase: Percentage of Participants With T-Cell Development
Description: Percentage of participants with T-Cell Development were planned to be reported.
Time Frame: From Week 188 up to end of study (Week 288)
Population: as for outcome 42
Arm/Group | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Group 1 and 2: Baseline up to Week 72 for participants who didn't enter LTE; up Week 216 for participants entering the LTE but not receiving late boost vaccination. Group 3: Baseline up to Week 72. Group 1b and 2b: From Week 188 up to Week 288.
Description: Groups 1 and 2: all randomized participants who received at least one dose in main study and continued in the LTE and did not enter late-boost vaccination phase; Group 3: all randomized participants and treated participants; Groups 1b and 2b: participants who received late-boost vaccination.
Arm/Group | Group 1 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 | Group 2 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 | Group 3 Main Study: Placebo | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine | Group 2b: LTE Then Late-boost Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/100 | 0/26 | 0/41 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/26 | 2/100 | 0/26 | 1/41 | 3/13
Other Adverse Events (participants affected / at risk) | 25/26 | 96/100 | 25/26 | 38/41 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 (N=26) | Group 2 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 (N=100) | Group 3 Main Study: Placebo (N=26) | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine (N=41) | Group 2b: LTE Then Late-boost Placebo (N=13)
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Death Neonatal (General disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Miscarriage of Partner (Social circumstances) | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 (N=26) | Group 2 Main Study and LTE Phase: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 (N=100) | Group 3 Main Study: Placebo (N=26) | Group 1b: LTE Then Late-boost Ad26.Mos4.HIV + gp140 HIV Bivalent Vaccine (N=41) | Group 2b: LTE Then Late-boost Placebo (N=13)
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Solicited) (Gastrointestinal disorders) | 9 | 46 | 9 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 6 | 0 | 0 | 0
Chills (Solicited) (General disorders) | 12 | 48 | 1 | 5 | 3
Erythema (Solicited) (General disorders) | 2 | 4 | 2 | 2 | 0
Fatigue (Solicited) (General disorders) | 19 | 78 | 18 | 26 | 7
Pain/Tenderness (Solicited) (General disorders) | 24 | 94 | 16 | 34 | 4
Pyrexia (Solicited) (General disorders) | 2 | 15 | 1 | 1 | 0
Swelling/Induration (Solicited) (General disorders) | 2 | 3 | 0 | 1 | 0
Vessel Puncture Site Pain (General disorders) | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 6 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 7 | 1 | 2 | 1
Rhinitis (Infections and infestations) | 2 | 4 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 16 | 6 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 1 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 4 | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 2 | 2 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 7 | 1 | 0 | 0
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 15 | 68 | 9 | 16 | 0
Headache (Nervous system disorders) | 1 | 7 | 1 | 1 | 0
Headache (Solicited) (Nervous system disorders) | 15 | 69 | 16 | 20 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to change in planned analysis, safety data for main study and LTE were combined for Groups 1 and 2 as LTE was a follow up for the participants who were in main study in Groups 1 and 2 and no intervention was given in LTE. As both phases involved the same participants in continued monitoring, the data reflects ongoing safety assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT02935686/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT02935686/SAP_001.pdf